CLINICAL TRIAL: NCT02008591
Title: Comparison of Epidural Labor Pain Relief Techniques on Maternal and Fetal Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P001927
Record Dates: First submitted 2013-11-26; First posted 2013-12-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Laboring Women Requesting Neuraxial Labor Analgesia
Keywords: Neuraxial Technique; Epidural Technique; Dural Puncture Epidural Technique; Combined Spinal Epidural Technique; Labor Analgesia; Obstetric

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with computer generated (Microsoft Excel 2015) assignment placed in sealed envelopes.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Anesthesiologist performing technique and bedside nurse instructed not to reveal randomization arm to the patient or study co-investigator who was waiting outside the room, and notified only after completion of the neuraxial placement protocol.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Epidural Technique (Active Comparator): Bupivacaine 0.125% with Fentanyl 2 mcg/mL, 15 mL load over 5 min
  Interventions: Procedure: Epidural Technique versus Dural Puncture Epidural Technique versus Combined Spinal Epidural Technique
- Combined Spinal Epidural Technique (Active Comparator): Bupivacaine 2.5 mg with Fentanyl 25 mcg
  Interventions: Procedure: Epidural Technique versus Dural Puncture Epidural Technique versus Combined Spinal Epidural Technique
- Dural Puncture Epidural Technique (Active Comparator): Bupivacaine 0.125% with Fentanyl 2 mcg/mL, 15 mL load over 5 min
  Interventions: Procedure: Epidural Technique versus Dural Puncture Epidural Technique versus Combined Spinal Epidural Technique

INTERVENTIONS:
Procedure: Epidural Technique versus Dural Puncture Epidural Technique versus Combined Spinal Epidural Technique — Three different techniques, using the same medications (bupivacaine and fentanyl)

SUMMARY:
The primary objective of this study is to compare the onset and duration of the initial dose of medications given through three different epidural (conventional epidural, combined spinal epidural and dural puncture epidural) techniques for labor pain relief.

The secondary objective of this study is to compare the fetal effects of these three epidural labor analgesia techniques.

ELIGIBILITY:
Inclusion Criteria:

* 1. Nulliparous (first baby) parturient 2. Singleton, vertex gestation at term (37-42 weeks) 3. Less than 5 cm dilation 4. Desires an epidural technique for labor analgesia

Exclusion Criteria:

- 1. Current or historical evidence of clinically significant disease or condition, including diseases of pregnancy (i.e preeclampsia, gestational diabetes) 2. Any contraindication to the administration of an epidural technique 3. History of hypersensitivity or idiosyncratic reaction to local anesthetic or opioid medications 4. Current or historical evidence of a disease which may result in the risk of a cesarean delivery.

5. Evidence of anticipated fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
Maternal Outcomes | Participants will be followed for the duration of labor analgesia from initiation to delivery, an expected average of 12 hours
  Onset, quality, and duration of analgesia, occurrences of hypotension, bradycardia, pruritus, nausea, emesis.

SECONDARY OUTCOMES:
Fetal Outcomes | Participants will be followed for the duration of labor analgesia from initiation to delivery, an expected average of 12 hours
  Occurrence of fetal bradycardia or other heart rate changes, changes in fetal heart tracing patterns

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Tsen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States